CLINICAL TRIAL: NCT00291200
Title: Enhancing the Prospective Prediction of Psychosis
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: MH61282; 5U01MH066160 (NIH); DATR AD-P
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Psychosis; Basic Symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for routine laboratory studies

GROUPS / COHORTS (2):
- 1: Participants with basic symptoms of psychosis
- 2: Control participants

SUMMARY:
This study will gather information on the natural history of the basic symptoms of psychosis to identify factors that may affect the improvement or persistence of the symptoms.

DETAILED DESCRIPTION:
Psychosis is a serious mental condition in which a person momentarily loses contact with reality. People in a state of psychosis may experience hallucinations or delusional beliefs that make day-to-day functioning difficult. During the early development of psychosis, people undergo an initial change in mood, thinking, or behavior that may include making mistakes about smells, sounds, or sights; becoming easily distracted; and developing suspicions of others. These basic symptoms can be early warning signs of a brain disorder, including anxiety disorder, depression, or psychotic disorder. Basic symptoms may be due to a number of factors, including a reaction to stress or drugs or just a part of normal adolescence. To identify psychosis early and accurately, more information is needed on the initial stages, biological markers, and progression of psychosis. This study will gather information on the natural history of the basic symptoms of psychosis to identify factors that may affect the improvement or persistence of the symptoms.

Participation in this study will last up to 5 years. The initial screening visit will be used to determine whether a participant is eligible for the group displaying basic symptoms or the control group. Initial screening will include giving a blood sample for routine lab tests, a physical exam, a drug test, and questions about medical history and symptoms. All participants will then partake in baseline evaluations, which involve assessments concerning concentration, problem solving, memory, social skills, and ability to identify smells. Participants will also respond to questions about symptoms, school and social functioning, stressful situations, and family history of illnesses. The participants who meet the criteria for basic symptoms will attend monthly 1-hour follow-up visits for the first year of the study. During these visits, participants will be asked about the status of their basic symptoms and use of medications. For the second year of the study, follow-up visits will occur every 2 months, and for the third, fourth, and fifth years of the study, visits will be every 3 months. Repeat baseline assessments will occur every 6 months, with each assessment visit lasting about 5 hours. All participants will undergo endpoint evaluations that follow the same format as most baseline assessments. Participants who develop a psychotic disorder during the study will attend an additional follow-up visit 6 months after the endpoint evaluation to confirm diagnosis. Participants who decide that they no longer wish to attend regular study visits may be asked to participate in follow-up telephone interviews about their basic symptoms every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets modified criteria of prodromal syndromes (COPS) for schizophrenia prodrome or help-seeking control

Exclusion Criteria:

* History of psychosis
* Antipsychotic treatment in the month prior to study entry
* More than 16 weeks of lifetime antipsychotic treatment

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of participants who meet the basic symptoms for psychosis and control participants recruited at three sites: the PRIME Clinics at University of North Carolina, Yale University, and the Center for Addiction and Mental Health (CAMH) in Toronto, Canada.
Sampling Method: Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2003-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Information on the natural history of basic symptoms of psychosis | Measured monthly during Year 1; every 2 months during Year 2; and every 3 months during Years 3, 4, and 5
Factors that may affect the improvement or persistence of basic symptoms of psychosis | Measured monthly during Year 1; every 2 months during Year 2; and every 3 months during Years 3, 4, and 5

CONTACTS AND LOCATIONS:
Overall Officials: Scott W. Woods, MD, Principal Investigator — Yale University; Jean Addington, PhD, Principal Investigator — University of Toronto; Diana O. Perkins, MD, MPH, Principal Investigator — University of North Carolina
Locations (3):
- United States (2):
  - Prevention through Risk Identification Management and Education (PRIME) Clinic, New Haven, Connecticut
  - PRIME Clinic, Chapel Hill, North Carolina
- PRIME Clinic, Toronto, Ontario, Canada